CLINICAL TRIAL: NCT05818475
Title: Functional Coronary Angiography to Indicate and Guide Revascularization in STEMI Patients with Multivessel Disease
Brief Title: Functional Coronary Angiography Guided Revascularization in STEMI
Acronym: AIR-STEMI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Simone Biscaglia, Study Principal Investigator, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 82/2023/Sper/AOUFe
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Myocardial Infarction
Keywords: Percutaneous coronary intervention; Angiography-derived Fractional Flow Reserve; Multivessel disease
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Independent Clinical Event Committee blinded to patient's arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Angiography-guided PCI (Active Comparator): Patients will receive PCI of all lesions with at least 50% diameter stenosis at visual estimation. PCI plan and assessment of PCI results will be based on angiography.
  Interventions: Other: Angiography-guided PCI
- Angiography-derived FFR PCI indication and planning (Experimental): Patients will receive PCI of all lesions with at least 50% diameter stenosis and positive angiography-derived FFR value (≤0.80). PCI planning will be based on the pullback curve obtained by angiography-derived FFR to obtain an optimal post-PCI physiology.
  Interventions: Other: Angiography-derived FFR PCI indication and planning

INTERVENTIONS:
Other: Angiography-guided PCI — Non-culprit lesion treatment will be based on visual estimation by angiography. The evaluation of PCI result will be also based only on angiography.
  Arms: Angiography-guided PCI
Other: Angiography-derived FFR PCI indication and planning — Non-culprit lesion treatment will be based on angiography-derived FFR result. In case of positive assessment, PCI will be planned according to the virtual PCI plan based on the physiology pullback curve.
  Arms: Angiography-derived FFR PCI indication and planning

SUMMARY:
The goal of this multicenter randomized clinical trial is to test the superiority in terms of efficacy of the Angiography-derived fractional flow reserve (AIR) over that based on conventional angiography (ANGIO) strategy in the management of non-culprit lesions in STEMI patients with multivessel disease.

The main questions it aims to answer are:

* is an Angiography-derived fractional flow reserve strategy superior to a conventional angiography strategy in reducing the occurrence of the composite efficacy endpoint of all-cause death, myocardial infarction, cerebrovascular accident, or ischemia-driven revascularization.
* is an Angiography-derived fractional flow reserve strategy superior to a conventional angiography strategy in reducing the occurrence of the composite safety endpoint of of contrast-associated acute kidney injury and Bleeding Academic Research Consortium (BARC) type 3-5.

Participants will be randomized after the successful treatment of the culprit lesion to one of the two strategies and prospectively followed-up.

DETAILED DESCRIPTION:
Reperfusion of the culprit lesion through primary PCI is the standard of care in ST-segment elevation myocardial infarction (STEMI) patients, regardless of their age. The actual gold standard for the management of non-culprit lesions in STEMI patients with multivessel disease (MVD) is angiography-guided complete revascularization. The Complete vs Culprit-only Revascularization to Treat Multi-vessel Disease after Primary PCI for STEMI (COMPLETE) trial randomized 4 041 patients with STEMI and MVD. The main finding was the highly significant reduction of new MI occurrence in the complete group (7.9% vs 5.4%, hazard ratio (HR) 0.68, 95% CI 0.53-0.87, p=0.002). Revascularization was obtained largely by angiographic evaluation (>99%).

After COMPLETE, the subsequent step was to ascertain which complete revascularization strategy should be pursued. In particular, physiology-guided revascularization was compared to an angio-guided strategy. The advantages of physiology against angiography are related to: a) lower number of vessels treated, b) lower number of stents implanted; c) avoidance of a second procedure in negative fractional flow reserve (FFR) patients during primary PCI; d) possibility to optimize the procedure from the physiological standpoint after percutaneous coronary intervention (PCI).

In the Flow Evaluation to Guide Revascularization in Multivessel ST-Elevation Myocardial Infarction (FLOWER-MI), patients with STEMI and multivessel disease who had undergone successful PCI of the infarct-related artery were randomly assigned to receive complete revascularization guided by either FFR or angiography. The primary outcome was a composite of death from any cause, nonfatal myocardial infarction, or unplanned hospitalization leading to urgent revascularization at 1 year. FFR-guided revascularization was associated with lower number of stents implanted per patient (1.01±0.99 versus 1.50±0.86). During follow-up, a primary outcome event occurred in 32 of 586 patients (5.5%) in the FFR-guided group and in 24 of 577 patients (4.2%) in the angiography-guided group (hazard ratio, 1.32; 95% confidence interval, 0.78 to 2.23; P = 0.31). Death occurred in 9 patients (1.5%) in the FFR-guided group and in 10 (1.7%) in the angiography-guided group; nonfatal myocardial infarction in 18 (3.1%) and 10 (1.7%), respectively; and unplanned hospitalization leading to urgent revascularization in 15 (2.6%) and 11 (1.9%), respectively.

The results of the FLOWER-MI trial may suggest that physiology can provide a similar outcome if compared to a conventional angio-guided approach. However, some limitation should be acknowledged: i) rate of events was three-times lower than expected suggesting both a selection bias and the need of a higher number of patients to demonstrate any difference among the two groups; ii) all patients in the FFR-group received a staged procedure to perform physiology assessment diluting one of the major advantages in FFR negative patients, namely the avoidance of a second procedure if physiology is negative; iii) in 16% of patients in the physio-guided group FFR was not performed before PCI, whereas in 82% of patients it was not performed after PCI; iv) even if FFR was associated with lower PCIs, periprocedural MI was three times higher if compared to the angio-group, suggesting its possible underreporting in the angio-group.

After the COMPLETE trial2, the actual standard of care in the management of STEMI patients with MVD is complete revascularization based on angiography. However, this approach may lead to over- or under-estimation of lesions in a relevant portion of patients with negative impact on prognosis. Invasive physiology has been consistently shown to be superior if compared to angio-guided strategy, but it is underutilized in clinical practice mainly due to feasibility issues.

A functional coronary angiography could overcome the applicability issues related to invasive physiology. In addition, it is particularly appealing in the evaluation of non-culprit lesions since:

1. It is possible to acquire projection during primary PCI and perform the analysis off-line
2. In case of negative assessment, the patient can avoid a second procedure to invasively measure physiology
3. It is possible to optimize most of the procedures by the physiological standpoint through the utilization of the virtual-PCI planner tool pre-PCI without the need to repeat physiology after PCI.
4. It has been recently shown that if compared to an angio-guided approach, Angiography-derived FFR was able to reduce the incidence of spontaneous MI by 36% Therefore, a strategy based on functional coronary angiography to indicate and guide PCI could be superior if compared to an angio-guided strategy both from the efficacy (CV death, cerebrovascular accident, MI and ischemia-driven revascularization) and from the safety (BARC 3-5, contrast-associated acute kidney injury) standpoint.

ELIGIBILITY:
Inclusion Criteria:

* ST-segment elevation myocardial infarction with indication to invasive management
* Multi-vessel disease defined as at least 1 non-culprit coronary artery lesion at least 2.5 mm in diameter deemed at visual estimation with a diameter stenosis % ranging from 50 to 99% amenable to successful treatment with PCI
* Successful treatment of culprit lesion

Exclusion Criteria:

* Planned surgical revascularization
* Left main as non-culprit lesion
* Non-cardiovascular co-morbidity reducing life expectancy to < 1 year
* Any factor precluding 1-year follow-up
* Prior Coronary Artery Bypass Graft (CABG) Surgery
* Impossibility to identify a clear culprit lesion
* Presence of a chronic total occlusion (CTO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1823 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Outcome: Patient Oriented Composite Outcome | through study completion, an average of 18 months
  Cumulative occurrence of mortality, cerebrovascular accident, reinfarction, or ischemia-driven revascularization
Primary Safety Outcome: Major Bleeding and Contrast - Associated Acute Kidney Injury | through study completion, an average of 18 months
  Cumulative occurrence of contrast-associated acute kidney injury and bleeding BARC 3-5

SECONDARY OUTCOMES:
Main Secondary Outcome: Cardiovascular Mortality and Myocardial Infarction | through study completion, an average of 18 months
  Cumulative occurrence of cardiovascular mortality and myocardial infarction

CONTACTS AND LOCATIONS:
Locations (22):
- Italy (21):
  - AUSL Bologna Ospedale Maggiore, Bologna, BO
  - Azienda Ospedaliero Universitaria di Ferrara, Ferrara, FE
  - Ospedale di Bolzano, Bolzano, Italy
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro, Italy
  - Ospedale Annunziata, Cosenza, Italy
  - Ospedale Civile di Baggiovara, Baggiovara, MO
  - AUSL Piacenza, Piacenza, PC
  - Azienda Ospedaliero Universitaria di Parma, Parma, PR
  - Arcispedale Santa Maria Nuova di Reggio Emilia, Reggio Emilia, RE
  - AUSL Romagna Ospedale degli Infermi Rimini, Rimini, RN
  - Ospedale Santa Maria della Misericordia Rovigo, Rovigo, RO
  - Ospedale dell'Angelo Mestre, Mestre, VE
  - Ospedale Mater Salutis Legnago, Legnago, VR
  - Azienda Ospedaliero Universitaria Integrata di Verona, Verona, VR
  - ASST Papa Giovanni XXIII, Bergamo
  - AORN Sant'Anna e San Sebastiano, Caserta
  - Ospedale Santa Maria Goretti, Latina
  - Ospedale Maggiore della Carità Novara, Novara
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - AUSL Romagna Santa Maria delle Croci Ravenna, Ravenna
  - Policlinico Casilino, Roma
- NICVD Karachi, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The present study is powered for the patient oriented composite endpoint, but not for CV death and MI. In order to obtain compelling evidence on this latter endpoint, the data of the present study will be merged with those of randomized clinical trials sharing the same inclusion and exclusion criteria, randomization and study interventions.
Supporting Information: Study Protocol
Time Frame: Data will be available for individual patient level analysis in order to merge our data with other trials sharing inclusion and exclusion criteria. Data will be available after the completion of the primary endpoint.
Access Criteria: Direct request to study Principal Investigator.

REFERENCES:
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Mehta SR, Wood DA, Cairns JA. Complete Revascularization with Multivessel PCI for Myocardial Infarction. Reply. N Engl J Med. 2020 Apr 16;382(16):1571-1572. doi: 10.1056/NEJMc2000278. No abstract available. PMID 32294360
- [Background] Pavasini R, Biscaglia S, Barbato E, Tebaldi M, Dudek D, Escaned J, Casella G, Santarelli A, Guiducci V, Gutierrez-Ibanes E, Di Pasquale G, Politi L, Saglietto A, D'Ascenzo F, Campo G. Complete revascularization reduces cardiovascular death in patients with ST-segment elevation myocardial infarction and multivessel disease: systematic review and meta-analysis of randomized clinical trials. Eur Heart J. 2020 Nov 7;41(42):4103-4110. doi: 10.1093/eurheartj/ehz896. PMID 31891653
- [Background] Collison D, Didagelos M, Aetesam-Ur-Rahman M, Copt S, McDade R, McCartney P, Ford TJ, McClure J, Lindsay M, Shaukat A, Rocchiccioli P, Brogan R, Watkins S, McEntegart M, Good R, Robertson K, O'Boyle P, Davie A, Khan A, Hood S, Eteiba H, Berry C, Oldroyd KG. Post-stenting fractional flow reserve vs coronary angiography for optimization of percutaneous coronary intervention (TARGET-FFR). Eur Heart J. 2021 Dec 1;42(45):4656-4668. doi: 10.1093/eurheartj/ehab449. PMID 34279606
- [Background] Biscaglia S, Uretsky B, Barbato E, Collet C, Onuma Y, Jeremias A, Tebaldi M, Hakeem A, Kogame N, Sonck J, Escaned J, Serruys PW, Stone GW, Campo G. Invasive Coronary Physiology After Stent Implantation: Another Step Toward Precision Medicine. JACC Cardiovasc Interv. 2021 Feb 8;14(3):237-246. doi: 10.1016/j.jcin.2020.10.055. PMID 33541534
- [Background] Biscaglia S, Tebaldi M, Brugaletta S, Cerrato E, Erriquez A, Passarini G, Ielasi A, Spitaleri G, Di Girolamo D, Mezzapelle G, Geraci S, Manfrini M, Pavasini R, Barbato E, Campo G. Prognostic Value of QFR Measured Immediately After Successful Stent Implantation: The International Multicenter Prospective HAWKEYE Study. JACC Cardiovasc Interv. 2019 Oct 28;12(20):2079-2088. doi: 10.1016/j.jcin.2019.06.003. Epub 2019 Sep 25. PMID 31563688
- [Background] Rioufol G, Derimay F, Roubille F, Perret T, Motreff P, Angoulvant D, Cottin Y, Meunier L, Cetran L, Cayla G, Harbaoui B, Wiedemann JY, Van Belle E, Pouillot C, Noirclerc N, Morelle JF, Soto FX, Caussin C, Bertrand B, Lefevre T, Dupouy P, Lesault PF, Albert F, Barthelemy O, Koning R, Leborgne L, Barnay P, Chapon P, Armero S, Lafont A, Piot C, Amaz C, Vaz B, Benyahya L, Varillon Y, Ovize M, Mewton N, Finet G; FUTURE Trial Investigators. Fractional Flow Reserve to Guide Treatment of Patients With Multivessel Coronary Artery Disease. J Am Coll Cardiol. 2021 Nov 9;78(19):1875-1885. doi: 10.1016/j.jacc.2021.08.061. PMID 34736563
- [Background] Puymirat E, Cayla G, Simon T, Steg PG, Montalescot G, Durand-Zaleski I, le Bras A, Gallet R, Khalife K, Morelle JF, Motreff P, Lemesle G, Dillinger JG, Lhermusier T, Silvain J, Roule V, Labeque JN, Range G, Ducrocq G, Cottin Y, Blanchard D, Charles Nelson A, De Bruyne B, Chatellier G, Danchin N; FLOWER-MI Study Investigators. Multivessel PCI Guided by FFR or Angiography for Myocardial Infarction. N Engl J Med. 2021 Jul 22;385(4):297-308. doi: 10.1056/NEJMoa2104650. Epub 2021 May 16. PMID 33999545
- [Background] Xu B, Tu S, Song L, Jin Z, Yu B, Fu G, Zhou Y, Wang J, Chen Y, Pu J, Chen L, Qu X, Yang J, Liu X, Guo L, Shen C, Zhang Y, Zhang Q, Pan H, Fu X, Liu J, Zhao Y, Escaned J, Wang Y, Fearon WF, Dou K, Kirtane AJ, Wu Y, Serruys PW, Yang W, Wijns W, Guan C, Leon MB, Qiao S, Stone GW; FAVOR III China study group. Angiographic quantitative flow ratio-guided coronary intervention (FAVOR III China): a multicentre, randomised, sham-controlled trial. Lancet. 2021 Dec 11;398(10317):2149-2159. doi: 10.1016/S0140-6736(21)02248-0. Epub 2021 Nov 4. PMID 34742368
- [Derived] Erriquez A, Colaiori I, Hakeem A, Guiducci V, Menozzi M, Barbierato M, Arioti M, D'Amario D, Casella G, Scarsini R, Polimeni A, Donazzan L, Benatti G, Venturi G, Ruozzi M, Giordan M, Monello A, Moretti F, Versaci F, Shah JA, Lakho AA, Mantovani F, Cavazza C, Bugani G, Lanzilotti V, Gallo F, Leone AM, Tebaldi M, Pavasini R, Piccolo R, Verardi FM, Farina J, Caglioni S, Cocco M, Campo G, Biscaglia S. Functional coronary angiography to indicate and guide revascularization in STEMI patients with multivessel disease: Rationale and design of the AIR-STEMI trial. Am Heart J. 2025 Jun;284:71-80. doi: 10.1016/j.ahj.2025.02.012. Epub 2025 Feb 19. PMID 39984150